CLINICAL TRIAL: NCT00986141
Title: Effect of Selective Laser Trabeculoplasty (SLT) on Diurnal Intraocular Pressure in Open-Angle Glaucoma Patients on Medical Treatment
Brief Title: Effects of Selective Laser Trabeculoplasty
Acronym: SLT
Status: Terminated | Type: Observational
Why Stopped: PI left the University
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 09-0315
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laser trabeculoplasty: Subjects with POAG and on medical treatment who are undergoing SLT
  Interventions: Procedure: Surgery; Procedure: Selective Laser Trabeculoplasty
- Surgery: Glaucoma laser treatment

INTERVENTIONS:
Procedure: Surgery — Selective Laser Trabeculoplasty for glaucoma
  Other Names: Selective Laser Trabeculoplasty
  Groups: laser trabeculoplasty
Procedure: Selective Laser Trabeculoplasty — Glaucoma Treatment
  Other Names: SLT
  Groups: laser trabeculoplasty

SUMMARY:
Primary objective is to evaluate the effect of selective laser trabeculoplasty (SLT) on the diurnal intraocular pressure variation in open-angle glaucoma patients (OAG).

DETAILED DESCRIPTION:
This is a prospective observational study of OAG patients undergoing selective laser trabeculoplasty at the University of Kentucky Chandler Medical Center. The patients will be recruited over 12 months. Study will include 3 visits: pre-laser visit, visit for laser treatment and post-laser visit. All visits will occur within a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have the diagnosis of open angle glaucoma
* Subjects who are able to speak and understand English and provide meaningful written informed consent,
* Subjects who are willing and able to comply with all testing and requirements defined in the protocol and willing and able to comply with all required study visits.

Exclusion Criteria:

* Subjects with previous laser treatment or intraocular surgery,
* Subjects with history of ocular inflammation and with history of previous ocular trauma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients, between the ages of 40 and 80, of either gender, from all ethnic backgrounds will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of selective laser trabeculoplasty on the diurnal intraocular pressure variation in OAG patients. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Davis, Assoc V Chair, Study Director — Univ of KY Reseach Foundation
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States